CLINICAL TRIAL: NCT00737061
Title: A Multi-Center, Prospective Evaluation of the Adiana System for Transcervical Sterilization Using Electrothermal Energy in Women Aged 18-45 - The EASE Trial
Brief Title: Safety & Efficacy Study of the Adiana System for Women Who Desire Permanent Birth Control (Sterilization)
Acronym: EASE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Product Pre-Market Approval withdrawn
Sponsor: Hologic, Inc. (Industry)
Collaborators: QST Consultations, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: P0071
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2013-01-25 (Estimated); Last update posted 2017-09-08 (Actual); Status verified 2017-08

CONDITIONS: Reproductive Sterilization
Keywords: Female; Sterilization

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Adiana Transcervical Sterilization System (Experimental): Single arm treatment
  Interventions: Device: Adiana Transcervical Sterilization System

INTERVENTIONS:
Device: Adiana Transcervical Sterilization System — Implantation of silicone matrix in fallopian tubes

SUMMARY:
The purpose of this study is to demonstrate the safety & efficacy of the Adiana Transcervical Sterilization System for women who desire permanent birth control (female sterilization) by occlusion of the fallopian tubes.

DETAILED DESCRIPTION:
Participants who demonstrated to be bilaterally occluded by hysterosalpingogram (HSG) evaluations are allowed to rely on the Adiana System for pregnancy prevention and enter the Wearing Period of follow-up.

Secondary endpoints inlcude safety of device placement procedure and safety of device wearing. The adverse events recorded during the course of the study are entered under adverse events.

ELIGIBILITY:
Inclusion Criteria:

* • Women aged 18 to 45

  * Women who are seeking permanent contraception
  * Women who are at risk of becoming pregnant
  * Willing to risk becoming pregnant when relying on the Adiana device for contraception
  * Relatively normal uterine cavity, uterine wall thickness, and uterine size as demonstrated by pelvic sonography
  * Willing to keep a coital/menstrual log
  * Have at least one confirmed pregnancy and one living child
  * Monogamous relationship with a partner who has proven fertility
  * Sexually active (at least 4 acts of intercourse per month)
  * Willing to use alternate contraception (either a barrier method or oral contraceptive pills or other monthly, cyclic, hormonal birth control) during the three months following device placement prior to relying on the Adiana device for contraception
  * Willing and able to maintain in regular contact with the investigator
  * Women with regular, cyclical menses within 2 months prior to the device placement procedure
  * Able to provide informed consent

Exclusion Criteria:

* Women who are unsure of their desire to end their fertility
* Presence of gross genital infection, including sepsis
* Presence of chlamydia, gonorrhea or syphilis
* Presence of genital cancer (note: CIN1 is acceptable)
* Intra-uterine pathology which would prevent optimal access to the tubal ostium and intramural portion of the fallopian tube, such as large submucous fibroids or uterine adhesions
* History of chronic pelvic pain (present within the previous year), prior ectopic pregnancy, or fallopian tube surgery, or currently diagnosed severe dysmenorrhea, severe dyspareunia, endometriosis, adenomyosis, or pelvic inflammatory disease
* Women with unresolved tubal, ovarian or endometrial pathology
* Uterine neoplasia or precursors to neoplasia
* Dysfunctional uterine bleeding or intermenstrual bleeding within the prior three months
* Women who have not had at least two normal periods after the following events: irregular periods treated with oral contraceptives (or other monthly, cyclic, hormonal birth control) which have since been discontinued, IUD removal, childbirth, or termination of pregnancy
* Currently taking immunosuppressive medications including steroids
* Pregnancy
* Uterine perforation within the last 3 months
* Contraindications for surgical methods of sterilization
* Less than three months have passed since the last delivery or abortion

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 770 (Actual)
Dates: Start 2002-11; Primary Completion 2005-12 (Actual); Study Completion 2013-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Evantash, MD, Study Director — Hologic, Inc.
Locations (16):
- United States (14):
  - Women's Health Research, Phoenix, Arizona
  - Kaiser Permanente, Roseville, California
  - Kaiser Permanente, San Rafael, California
  - Reproductive Science Center, San Ramon, California
  - Center for Fertility and Women's Health, New Britain, Connecticut
  - Institute for Women's Health and Body, Wellington, Florida
  - Center for Reproductive Medicine, Wichita, Kansas
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Minnesota Gynecology and Surgery, Edina, Minnesota
  - St. Luke's Hospital, Chesterfield, Missouri
  - Duke Fertility Center, Durham, North Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Fort Worth, Texas
  - Reproductive Specialty Center, Milwaukee, Wisconsin
- Royal Hospital for Women, Randwick, New South Wales, Australia
- Hospital Universitario UANL, Monterrey, Nuevo León, Mexico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled in the trial from 16 investigative sites between November 13, 2002 and April 28, 2005. Fourteen sites were located in the US and two were international sites.
Pre-assignment Details: 770 subjects were enrolled: 75 withdrew consent and 50 were excluded for pathology/procedural criteria. All subjects were enrolled on an intent to treat (ITT) basis. The ITT population included all patients who were enrolled in the study and had device placement attempted. 645 subjects had treatment attempted. No comparative assessment was made.
Groups:
- Adiana Permanent Contraception System: Implantation of silicone matrix in fallopian tubes
Period: Waiting Period
Arm/Group | Adiana Permanent Contraception System
Started | 645
Completed | 570
Not Completed | 75
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 1
Not completed — Bilateral placement failure | 34
Not completed — Deemed patent following HSG | 26
Not completed — Alternative contraception failure | 3
Not completed — Elected surgical tubal ligation | 5
Period: 1 Year Wearing Period
Arm/Group | Adiana Permanent Contraception System
Started | 570
Completed | 553
Not Completed | 17
Not completed — Lost to Follow-up | 11
Not completed — Withdrawal by Subject | 2
Not completed — Discontinued reilance | 3
Not completed — Terminated for protocol non-compliance | 1

BASELINE CHARACTERISTICS:
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 645
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 645
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years]
  All Participants | 31.5 [20 to 45]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 645
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: 1 Year Pregnancy Rate
Description: Pregnancy rate is defined as the cumulative percentage of pregnancies occuring within the time frame. The primary endpoint for this study is the pregnancy prevention rate after one year of reliance on the Adiana System for pregnancy prevention. The pregnancy rate was evaluated for all participants who underwent successful bilateral treatment and who had demonstrated tubal occlusion by hysterosalpingogram (HSG) at the end of the Waiting Period.
Time Frame: 1 year
Population: 645 participants had treatment attempted; Intent to Treat population. Of these 645, 570 were able to rely on the device and are used to evaluate the pregnancy prevention rate for the 1-year endpoint. During the 1-year follow-up period, there were 6 pregnancies, of which 3 were attributable to physician error, i.e., misinterpretation of HSG results.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 570
percentage of participants | 1.1
Statistical Analysis 1: Comparison: Adiana Permanent Contraception System; 1-sided confidence interval. No statistical hypothesis testing was performed. Confidence interval represents a 1-sided confidence interval for the pregnancy prevention rate in the EASE Trial. 95% confidence interval derived using Kaplan Meier methods (log-log with PETO adjustment); Test type: Superiority or Other; Pregnancy Prevention Rate = 98.9, 95% CI [97.9 to 100]
Statistical Analysis 2: Comparison: Adiana Permanent Contraception System; 2-sided confidence interval. No statistical hypothesis testing was performed. Confidence interval represents a 2-sided confidence interval for the pregnancy prevention rate in the EASE Trial. 95% confidence interval derived using Kaplan Meier methods (log-log with PETO adjustment); Test type: Superiority or Other; Pregnancy Prevention Rate = 98.9, 95% CI [97.6 to 99.5]

2. Secondary Outcome: Device Placement Rate
Description: Defined as successful bilateral tubal access followed by successful bilateral RF treatment and matrix placement.
Time Frame: After First Treatment Attempt
Population: Device placement rate reported on a per participant basis for 645 intent to treat participants. Successful bilateral placement of the matrices was achieved in 604/645 participants after the first procedure.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 645
percentage of participants | 93.6

3. Secondary Outcome: Device Placement Rate
Description: Defined as successful bilateral tubal access followed by successful bilateral RF treatment and matrix placement.
Time Frame: Including Second Treatment Attempt
Population: Device placement rate reported on a per participant basis for 645 intent to treat participants. Successful bilateral placement of the matrices was achieved in 611/645 participants after 7 participants underwent a successful second attempt.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 645
percentage of participants | 94.7

4. Secondary Outcome: Patient Satisfaction With Placement Procedure
Description: Determined by verbal questions up to 48 hours post placement. Endpoint reported represents minimum percentage of participants reporting somewhat satisfied, satisfied or very satisfied.
Time Frame: 48 hours
Population: Intent to treat population; no imputations for missing data. Minimum satisfaction reported as 605/625 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 625
percentage of participants | 96.8

5. Secondary Outcome: Patient Satisfaction With Device Wearing
Description: Determined by verbal questions during periodic follow-up contacts. Endpoint reported represents minimum percentage of subjects reporting somewhat satisfied, satisfied or very satisfied.
Time Frame: Waiting Period (1-Month, 2-Months, 3-Months)
Population: Intent to treat population; no imputations for missing data. Minimum satisfaction reported at 2-Months as 587/613 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 613
percentage of participants | 95.8

6. Secondary Outcome: Patient Satisfaction With Device Wearing
Description: as for outcome 5
Time Frame: Wearing Period (3-Months, 6-Months, 9-Months, 12-Months)
Population: Per protocol population; no imputations for missing data. Minimum satisfaction reported at 12-Months as 528/531 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 531
percentage of participants | 99.4

7. Secondary Outcome: Patient Comfort With Placement Procedure
Description: Determined by verbal questions two hours following procedure or at discharge from facility, whichever came first. Endpoint reported represents minimum percentage of participants reporting any discomfort or pain experienced during the procedure as the same as or less than they expected.
Time Frame: Post-Procedure
Population: Intent to treat population; no imputations for missing data. Minimum comfort reported as 504/629 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 629
percentage of participants | 80.1

8. Secondary Outcome: Patient Comfort With Placement Procedure
Description: Determined by verbal questions up to 48 hours post placement. Endpoint reported represents minimum percentage of participants reporting any discomfort or pain experienced in first 48 hours following procedure as the same as they expected, less than they expected or no pain.
Time Frame: 48 hours
Population: Intent to treat population; no imputations for missing data. Minimum comfort reported as 578/632 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 632
percentage of participants | 91.5

9. Secondary Outcome: Patient Comfort With Device Wearing
Description: Determined by verbal questions during periodic follow-up contacts. Endpoint represents minimum percentage of subjects reporting good, very good or excellent comfort.
Time Frame: Waiting Period (1-Month, 2-Months, 3-Months)
Population: Intent to treat population; no imputations for missing data. Minimum comfort reported at 1-Month as 604/608 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 608
percentage of participants | 99.3

10. Secondary Outcome: Patient Comfort With Device Wearing
Description: as for outcome 9
Time Frame: Wearing Period (3-Months, 6-Months, 9-Months, 12-Months)
Population: Per protocol population; no imputations for missing data. Minimum comfort reported at 12-Months as 530/532 participants.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 532
percentage of participants | 99.6

11. Secondary Outcome: 3 Year Pregnancy Rate
Description: Pregnancy rate is defined as the cumulative percentage of pregnancies occuring within the time frame. The pregnancy rate was evaluated for all participants who underwent successful bilateral treatment and who had demonstrated tubal occlusion by hysterosalpingogram (HSG) at the end of the Waiting Period who have been followed for up to 3 years.
Time Frame: 3 years
Population: Population includes all participants able to rely on Adiana (n=570). This analysis is cumulative and based on survival analysis methodology. Thus, participants only followed for 2 years, for example, would still be included in this cumulative analysis. In total, 481 participants were available with 3 years of follow-up at the time of analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Adiana Permanent Contraception System
Number analyzed (Participants) | 570
percentage of participants | 1.6
Statistical Analysis 1: Comparison: Adiana Permanent Contraception System; 1-sided Confidence Interval. No hypothesis testing was performed. Confidence interval represents a 1-sided confidence interval for the pregnancy prevention rate in the EASE trial. 95% confidence interval derived using Kaplan Meier methods (log-log with PETO adjustment); Test type: Superiority or Other; No statistical hypothesis testing was performed; Pregnancy Prevention Rate = 98.4, 95% CI [97.2 to 100]
Statistical Analysis 2: Comparison: Adiana Permanent Contraception System; 2-sided Confidence Interval No hypothesis testing was performed. Confidence interval represents a 2-sided confidence interval for the pregnancy prevention rate in the EASE trial. 95% confidence interval derived using Kaplan Meier methods (log-log with PETO adjustment); Test type: Superiority or Other; No statistical hypothesis testing was performed; Pregnancy Prevention Rate = 98.4, 95% CI [96.9 to 99.1]

ADVERSE EVENTS:
Time Frame: Post-procedure, 48-Hours, 1-Week, 1-Month, 2-Months, 3-Months (Waiting Period), 3-Months (Wearing Period), participant diary through the 3-Month Wearing Period, 6-Months, 9-Months, 12-Months, 18-Months, 24-Months, 36-Months.
Description: Questions were asked through the 12-Month visit to assess subjects' presence or absence of post-operative discomfort. Subjects completed a participant diary detailing menstrual and sexual activity, and any symptoms, through the 3-Month Wearing Period. Follow-up visits included an assessment of subjects' potential adverse events.
Arm/Group | Adiana Permanent Contraception System
Serious Adverse Events (participants affected / at risk) | 60/645
Other Adverse Events (participants affected / at risk) | 642/645
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adiana Permanent Contraception System (N=645)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Basedow's disease (Endocrine disorders) | 1 (1)
Keratoconjunctivitis sicca (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Breast abscess (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 3 (3)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament injury (Injury, poisoning and procedural complications) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 1 (1)
Nerve injury (Injury, poisoning and procedural complications) | 1 (1)
Pain trauma activated (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Benign neoplasm of spinal cord (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 (4)
Monoplegia (Nervous system disorders) | 1 (1)
Multiple sclerosis (Nervous system disorders) | 2 (2)
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 2 (2)
Bipolar disorder (Psychiatric disorders) | 2 (2)
Depression (Psychiatric disorders) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Renal pain (Renal and urinary disorders) | 1 (1)
Adenomyosis (Reproductive system and breast disorders) | 2 (2)
Cervical dysplasia (Reproductive system and breast disorders) | 1 (1)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 2 (2)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 2 (2)
Ovarian cyst (Reproductive system and breast disorders) | 2 (2)
Pelvic pain (Reproductive system and breast disorders) | 3 (3)
Uterine polyp (Reproductive system and breast disorders) | 2 (2)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Gastric bypass (Surgical and medical procedures) | 3 (3)
Hernia hiatus repair (Surgical and medical procedures) | 1 (1)
Hysterectomy (Surgical and medical procedures) | 1 (1)
Mastectomy (Surgical and medical procedures) | 1 (1)
Surgery (Surgical and medical procedures) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adiana Permanent Contraception System (N=645)
Abdominal distension (Gastrointestinal disorders) | 55 (76)
Abdominal pain (Gastrointestinal disorders) | 51 (82)
Diarrhoea (Gastrointestinal disorders) | 35 (40)
Nausea (Gastrointestinal disorders) | 199 (270)
Vomiting (Gastrointestinal disorders) | 74 (89)
Hypersensitivity (Immune system disorders) | 44 (118)
Influenza (Infections and infestations) | 78 (90)
Nasopharyngitis (Infections and infestations) | 90 (115)
Sinusitis (Infections and infestations) | 59 (73)
Upper respiratory tract infection (Infections and infestations) | 38 (44)
Urinary tract infection (Infections and infestations) | 65 (78)
Vaginal mycosis (Infections and infestations) | 43 (58)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 34 (36)
Post procedural pain (Injury, poisoning and procedural complications) | 91 (118)
Arthralgia (Musculoskeletal and connective tissue disorders) | 116 (178)
Back pain (Musculoskeletal and connective tissue disorders) | 385 (1139)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 485 (895)
Neck pain (Musculoskeletal and connective tissue disorders) | 47 (76)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 (61)
Headache (Nervous system disorders) | 428 (2006)
Migraine (Nervous system disorders) | 70 (241)
Sinus headache (Nervous system disorders) | 42 (83)
Depression (Psychiatric disorders) | 59 (62)
Insomnia (Psychiatric disorders) | 36 (49)
Dysuria (Renal and urinary disorders) | 75 (83)
Amenorrhoea (Reproductive system and breast disorders) | 36 (51)
Dysmenorrhoea (Reproductive system and breast disorders) | 520 (2860)
Dyspareunia (Reproductive system and breast disorders) | 101 (186)
Menorrhagia (Reproductive system and breast disorders) | 146 (269)
Menstruation irregular (Reproductive system and breast disorders) | 52 (66)
Metrorrhagia (Reproductive system and breast disorders) | 573 (1149)
Muscle cramp (Reproductive system and breast disorders) | 72 (76)
Pelvic pain (Reproductive system and breast disorders) | 346 (924)
Polymenorrhoea (Reproductive system and breast disorders) | 33 (42)
Post procedural haemorrhage (Reproductive system and breast disorders) | 188 (208)
Vaginal discharge (Reproductive system and breast disorders) | 284 (738)
Vaginal haemorrhage (Reproductive system and breast disorders) | 255 (515)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 38 (44)

LIMITATIONS AND CAVEATS:
At the time of analysis, 481 completed 3 years. Due to the cumulative nature of the analysis, subjects may be lost to follow-up at one time and return to follow-up at a subsequent point. All subjects who have not withdrawn consent will be followed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All publications must be submitted for review and approval at least (30) days before the date on which it is to be submitted.

No publication of data wil be permitted prior to the submission and publication of the entire clinical trial.